CLINICAL TRIAL: NCT03945903
Title: SIMPONI SC Managed Access Program
Brief Title: Pre-Approval Access to Golimumab Subcutaneous for the Treatment of Stage 3 Type-1 Diabetes Mellitus in Children and Young Adults
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108621; CNTO148DML4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-04-24; First posted 2019-05-10 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — golimumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Golimumab — Participants will receive subcutaneous (SC) golimumab, where doses will be based on weight and/or body surface area.
  Other Names: SIMPONI

SUMMARY:
This is a Single Patient Investigational New Drug (IND) to golimumab subcutaneous (SC) for the treatment of recently diagnosed Stage 3 type-1 diabetes mellitus (T1D) in children and young adults. The main purpose of a single patient IND is to provide treatment to participants with serious/life-threatening diseases or conditions prior to marketing authorization.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Rady Children's Hospital, San Diego, California, United States